CLINICAL TRIAL: NCT04088357
Title: A Phase II, Closed Label, Randomized, Double Blind Study for the Treatment of Acute Induced Wounds With TolaSure Gel, 5% w/w in Healthy Volunteers
Brief Title: Efficacy of Topical TolaSure on Acute Induced Wounds in Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMendics, LLC (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYM 2019-01
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-06

CONDITIONS: Wound Healing
Keywords: Healthy Participants; Skin; Dermal; Biopsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 Percent TolaSure Topical Gel (Active Comparator): 5%(w/w) TolaSure Gel
  Interventions: Drug: TolaSure Topical Gel
- Topical Vehicle Gel (Placebo Comparator): Vehicle Gel
  Interventions: Drug: Topical Vehicle Gel

INTERVENTIONS:
Drug: TolaSure Topical Gel — TolaSure topical gel is applied to skin punch biopsies daily for the first seven consecutive days, then three times a week, defined as every two to three days, until closure.
  Other Names: Active Ingredient BM-3103
  Arms: 5 Percent TolaSure Topical Gel
Drug: Topical Vehicle Gel — TolaSure Vehicle Gel is applied topically to skin punch biopsies daily for the first seven consecutive days, then three times a week, defined as every two to three days, until closure.
  Other Names: TolaSure Vehicle Gel
  Arms: Topical Vehicle Gel

SUMMARY:
TolaSure is a topical gel for the promotion of accelerated wound healing. This phase II study will primarily assess the efficacy of TolaSure when applied to skin wounds created by punch biopsy in healthy participants. Safety, cutaneous tolerability, wound pain control, and quality of healing will also be assessed. A total of 80 healthy volunteers, males and females ages 18 years or older, will be enrolled. Subjects will be monitored for safety and efficacy until wound closure (estimation about 8 weeks) following topical administration of TolaSure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females > 18 years of age
* Health history review
* Physical exam
* Blood and urine clinical chemistries
* Negative pregnancy test

Exclusion Criteria:

* Acute or chronic skin disorders (e.g. psoriasis);
* Acne or dermatitis at the test site;
* Prone to keloids or hypertrophic scarring;
* Topical or systemic antibiotics within 4 weeks of study enrollment;
* Subjects with known severe mental illness which, in the investigator's opinion, may prevent informed consent or interfere with the subject's ability to comply with study protocol procedures;
* Diagnosed with Diabetes Type I/II or glucose results indicative of prediabetic condition;
* Morbidly obese with a Body Mass Index (BMI) ≥ 40;
* Surgery within the previous 3 months (except for minor cosmetic or dental procedures)
* History of severe vitamin or mineral deficiency;
* History of drug or alcohol abuse (as defined by the Investigator);
* Smoking/Vaping;
* HIV/AIDS;
* Consistently taking steroids and/or non-steroidal anti-inflammatory drugs. Subjects may use NSAIDs on an as needed basis with no more than 7 days of consecutive use;
* Cancer diagnosis in the last 5 years;
* Currently receiving chemotherapy or radiation;
* Women who are pregnant, nursing, or planning a pregnancy;
* Hyper- or hypo-pigmentation, or tattoos in the area where they will place the test fields;
* Symptoms of a clinically significant illness in the four weeks before treatment application that may influence the outcome of the study;
* Treatment with any investigational agent within one month before treatment application for this trial;
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule;
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Accelerated Wound Closure | Day 1, 2, and 7, then weekly until closure (estimated 8 weeks)
  Time-to-closure will be calculated by the number of days from biopsy to wound closure. Wound closure (changes in wound area (mm^2) over time) will be determined by the digital imaging platform software with Principal Investigator confirmation.

SECONDARY OUTCOMES:
Percent Area Reduction after Four Weeks | Week 4
  Wound area measurements (mm^2) will be calculated at week 4 by using a digital imaging. A percent reduction in area at week 4 will be calculated by comparing the initial area of the biopsy at Day 1 to the week 4 biopsy area.
Wound Pain Control | Day 2 and 7, then weekly until wound closure (estimated 8 weeks)
  Wound-related pain or discomfort will be assessed, using the Visual Analog Scale (VAS) for Pain, for each individual wound site as pain at rest followed by pain to touch.
  The VAS Pain is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length.
  Pain will be defined per the following scale:
  None - 0-4 mm; Mild - 5-44 mm: Moderate - 45-74; Severe - 75-100 mm
Quality of Healing | End of study (estimated 8 weeks)
  Patient and Observer Scar Assessment Scale (POSAS) version 2.0 will be used to assess the quality of healing of each biopsy site at the end of the study once both wounds are closed.
Cutaneous Tolerability | Day 1, 2, and 7, then weekly until wound closure (estimated 8 weeks)
  Cutaneous tolerability will include an evaluation of erythema and edema following the modified Draize scoring system. Draize scores will be recorded and changes from baseline Draize scores will be monitored over the course of the time frame.
  Draize Scoring System. Erythema: 0-No Erythema, 1-Slight Erythema, 2-Well Defined Erythema, 3- Moderate or Severe Erythema, 4- Severe Erythema or slight eschar formation.
  Edema: 0- No Edema, 1- Very Slight Edema(barely perceptible), 2-Slight Edema (well defined edges), 3-Moderate Edema (raised >1mm), 4- Severe Edema (raised >1mm and extending beyond the area of exposure)
Blood and Urine Chemistries | Screening, Day 2 and 7, then weekly until wound closure (estimated 8 weeks)
  Absolute values and changes over time of clinical chemistries including; Absolute values and changes over time of clinical blood and urine chemistries including; Hematology and Coagulation, Coagulation, Serum Chemistry, and Urinalysis. Blood and urine analytes are measured on a per mL basis.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - J&S Studies, College Station, Texas

IPD SHARING:
Plan to Share IPD: No